CLINICAL TRIAL: NCT07153991
Title: Efficacy of Donepezil in Patients With Chronic Tinnitus
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Elaine Miwa Watanabe, medical doctor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE 34251320.5.0000.0068; U1111-1248-6988 (Registry Identifier: UTN Universal Trial Number)
Record Dates: First submitted 2025-08-20; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Tinnitus
Keywords: tinnitus; donepezil
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention Group (donepezil) (Experimental): 35 Participants with tinnitus received donepezil for 3 months, starting with 5 mg daily for the first month and 10 mg daily for the following two months.
  Interventions: Drug: Donepezil group
- Placebo group (Placebo Comparator): 35 Pacients with tinnitus received for 3 months placebo medication
  Interventions: Drug: Placebo group

INTERVENTIONS:
Drug: Donepezil group — Participants received donepezil for 3 months, starting with 5 mg daily for the first month and 10 mg daily for the following two months
  Arms: Intervention Group (donepezil)
Drug: Placebo group — 35 Pacients with tinnitus received for 3 months placebo medication
  Arms: Placebo group

SUMMARY:
This study is a prospective, placebo-controlled, randomized, double-blind clinical trial, including 70 patients with chronic sensorineural tinnitus, divided into placebo and treatment groups. Participants received donepezil for 3 months, starting with 5 mg daily for the first month and 10 mg daily for the following two months.

DETAILED DESCRIPTION:
Treatment effects were monitored using the Tinnitus Handicap Inventory (THI) and the Visual Analogue Scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic sensorineural tinnitus type

Exclusion Criteria:

* pregnancy, arrhythmia, donepezil allergy, yelow dye allergy, otitis or any ear inflamatory diseases, patients taking any medication for dementia, convulsive diseases, asthma, patients taking any of these medications: carbamazepine, dexamethasone, phenobarbital, phenytoin, rifampicin, ketoconazole, quinidine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-11-19 (Actual); Primary Completion 2025-12-09 (Estimated); Study Completion 2025-12-09 (Estimated)

PRIMARY OUTCOMES:
tinnitus improvement | 3 months
  Treatment effects were monitored using the Tinnitus Handicap Inventory (THI) and the Visual Analogue Scale (VAS).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade De São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided